CLINICAL TRIAL: NCT00197041
Title: A Study to Evaluate the Safety, Immunogenicity and Efficacy of GlaxoSmithKline Biologicals' Candidate Malaria Vaccine RTS,S/AS02A, Administered Intramuscularly According to a 0, 1 and 2 Month Vaccination Schedule in Toddlers and Children Aged 1 to 4 Years in a Malaria-endemic Region of Mozambique.
Brief Title: A Study to Evaluate the Safety, Immunogenicity and Efficacy of GlaxoSmithKline (GSK) Biologicals' Candidate Malaria Vaccine RTS,S/AS02A, When Administered to Children Aged 1 to 4 Years Living in a Malaria-endemic Region of Mozambique.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 257049/026
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2016-09-21 (Estimated); Status verified 2016-09

CONDITIONS: Malaria
MeSH Terms: conditions — Malaria | interventions — RTS,S-AS02A vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

INTERVENTIONS:
Biological: RTS,S/AS02A

SUMMARY:
Malaria is an important cause of death and serious illness among Mozambican children. Although the risk of malaria can be reduced by drugs and by impregnated bed nets, it would be helpful if children could be protected against malaria by a vaccine.

GSK Biologicals is developing in partnership with Malaria Vaccine Initiative at PATH a candidate malaria vaccine RTS,S/AS02 for the routine immunization of infants and children living in malaria endemic areas. The vaccine would offer protection against malaria disease due to the parasite Plasmodium falciparum and also would provide protection against infection with hepatitis B virus. Previous studies have shown the candidate malaria vaccine RTS,S/AS02 to be safe when administered in adults and children aged 1-11 years. However, to assess if this vaccine could provide protection against malaria in children, this study has been undertaken.

DETAILED DESCRIPTION:
In this study, the participating children will either receive either 3 doses of the new malaria vaccine or the control vaccine which has been selected because of its benefit to the children in preventing important childhood diseases. The control vaccines include the following:

* If the child is of 24 months or older, he/she may receive 3 doses of a vaccine, called Engerix-B™, which protects against hepatitis B.
* If the child is less than 24 months, he/she may receive: two doses of a vaccine called Prevnar® and one dose of a vaccine called Hiberix™. Prevnar® prevents pneumonia and meningitis caused by some Streptococcus pneumoniae bacteria. Hiberix™ prevents severe infections such as pneumonia and meningitis caused by Haemophilus influenzae type b bacteria (Hib). All children will be monitored for the development of malaria disease over an 18-month period extending from the third vaccination. All participants will also be monitored for vaccine safety from first vaccination to study close.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female children, 1 to 4 years of age at the time of first vaccination (up to but not including 5th birthday).
* Written/thumbprinted and witnessed informed consent obtained from the parents or legal guardians.

Exclusion Criteria:

* Major congenital defects or serious chronic illness.
* History of allergic reactions to vaccination or to any component of the Hiberix™, Prevnar® or Engerix-B™ vaccines.
* Chronic administration (defined as more than 14 days) of immuno-suppressants or other immune modifying drugs within six months prior to the first vaccine dose .
* Previous vaccination with an experimental vaccine or with hepatitis B vaccine in children equal to or more than 18 months of age.
* Simultaneous participation in any other clinical trial.
* Use of any investigational or non-registered drug or vaccine other than the study vaccine(s) within 30 days preceding the first dose of study vaccine, or planned use during the study period.
* Planned administration of a vaccine not foreseen by the study protocol within 30 days before the first dose of vaccine. An exception, is the receipt of an EPI or licensed vaccine.
* Administration of immunoglobulins and/or any blood products within the three months preceding the first dose of study vaccine or planned administration during the study period.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, including human immunodeficiency virus (HIV) infection.

Ages: 1 Year to 4 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 2022 (Actual)
Dates: Start 2003-07; Primary Completion 2005-04 (Actual); Study Completion 2005-04 (Actual)

PRIMARY OUTCOMES:
Time to the first clinical episode of symptomatic Plasmodium falciparum malaria infection detected over the 6-month surveillance period after Dose 3 vaccination.

SECONDARY OUTCOMES:
Occurrence of episodes of asymptomatic and symptomatic infections of Plasmodium falciparum malaria. Occurrence of solicited symptoms, unsolicited symptoms and SAEs.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Maputo, Mozambique

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Jairoce C, Macia D, Torres-Yaguana JP, Mayer L, Vidal M, Santano R, Hurtado-Guerrero R, Reiter K, Narum DL, Lopez-Gutierrez B, Hamerly T, Sacarlal J, Aguilar R, Dinglasan RR, Moncunill G, Izquierdo L, Dobano C. RTS,S/AS02A Malaria Vaccine-Induced IgG Responses Equally Recognize Native-Like Fucosylated and Nonfucosylated Plasmodium falciparum Circumsporozoite Proteins. J Infect Dis. 2024 Mar 14;229(3):795-799. doi: 10.1093/infdis/jiad471. PMID 37889513
- [Derived] Feng G, Kurtovic L, Agius PA, Aitken EH, Sacarlal J, Wines BD, Hogarth PM, Rogerson SJ, Fowkes FJI, Dobano C, Beeson JG. Induction, decay, and determinants of functional antibodies following vaccination with the RTS,S malaria vaccine in young children. BMC Med. 2022 Aug 25;20(1):289. doi: 10.1186/s12916-022-02466-2. PMID 36002841
- [Derived] Cheung YB, Ma X, Lam KF, Milligan P. Estimation of the primary, secondary and composite effects of malaria vaccines using data on multiple clinical malaria episodes. Vaccine. 2020 Jul 6;38(32):4964-4969. doi: 10.1016/j.vaccine.2020.05.086. Epub 2020 Jun 12. PMID 32536547
- [Derived] Campo JJ, Dobano C, Sacarlal J, Guinovart C, Mayor A, Angov E, Dutta S, Chitnis C, Macete E, Aponte JJ, Alonso PL. Impact of the RTS,S malaria vaccine candidate on naturally acquired antibody responses to multiple asexual blood stage antigens. PLoS One. 2011;6(10):e25779. doi: 10.1371/journal.pone.0025779. Epub 2011 Oct 12. PMID 22022448
- [Derived] Aide P, Dobano C, Sacarlal J, Aponte JJ, Mandomando I, Guinovart C, Bassat Q, Renom M, Puyol L, Macete E, Herreros E, Leach A, Dubois MC, Demoitie MA, Lievens M, Vekemans J, Loucq C, Ballou WR, Cohen J, Alonso PL. Four year immunogenicity of the RTS,S/AS02(A) malaria vaccine in Mozambican children during a phase IIb trial. Vaccine. 2011 Aug 11;29(35):6059-67. doi: 10.1016/j.vaccine.2011.03.041. Epub 2011 Apr 7. PMID 21443960
- [Derived] Sacarlal J, Aide P, Aponte JJ, Renom M, Leach A, Mandomando I, Lievens M, Bassat Q, Lafuente S, Macete E, Vekemans J, Guinovart C, Sigauque B, Sillman M, Milman J, Dubois MC, Demoitie MA, Thonnard J, Menendez C, Ballou WR, Cohen J, Alonso PL. Long-term safety and efficacy of the RTS,S/AS02A malaria vaccine in Mozambican children. J Infect Dis. 2009 Aug 1;200(3):329-36. doi: 10.1086/600119. PMID 19569964
- [Derived] Guinovart C, Aponte JJ, Sacarlal J, Aide P, Leach A, Bassat Q, Macete E, Dobano C, Lievens M, Loucq C, Ballou WR, Cohen J, Alonso PL. Insights into long-lasting protection induced by RTS,S/AS02A malaria vaccine: further results from a phase IIb trial in Mozambican children. PLoS One. 2009;4(4):e5165. doi: 10.1371/journal.pone.0005165. Epub 2009 Apr 14. PMID 19365567
- [Derived] Alonso PL, Sacarlal J, Aponte JJ, Leach A, Macete E, Aide P, Sigauque B, Milman J, Mandomando I, Bassat Q, Guinovart C, Espasa M, Corachan S, Lievens M, Navia MM, Dubois MC, Menendez C, Dubovsky F, Cohen J, Thompson R, Ballou WR. Duration of protection with RTS,S/AS02A malaria vaccine in prevention of Plasmodium falciparum disease in Mozambican children: single-blind extended follow-up of a randomised controlled trial. Lancet. 2005 Dec 10;366(9502):2012-8. doi: 10.1016/S0140-6736(05)67669-6. PMID 16338450
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Annotated Case Report Form: 257049/026 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 257049/026 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 257049/026 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 257049/026 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 257049/026 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 257049/026 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 257049/026 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register